CLINICAL TRIAL: NCT03332173
Title: A Phase 2, Single-Arm, Open-Label, Multicenter Study of Bruton's Tyrosine Kinase (BTK) Inhibitor BGB-3111 in Chinese Subjects With Relapsed/Refractory Waldenström's Macroglobulinemia (WM)
Brief Title: Study of BTK Inhibitor BGB-3111 in Chinese Subjects With Relapsed/Refractory Waldenström's Macroglobulinemia (WM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-210; CTR20170208 (Registry Identifier: Center for drug evaluation, NMPA)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Waldenström's Macroglobulinemia (WM)
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Zanubrutinib 160 mg orally twice daily with or without food until progressive disease or intolerable toxicity
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Oral administration using 80 mg capsules
  Other Names: BGB-3111; Brukinsa

SUMMARY:
This was a single-arm, multicenter Phase 2 study in Chinese participants with relapsed or refractory Waldenström's macroglobulinemia who exhibited one or more of the criteria for requiring treatment based on consensus guidelines from the Seventh International Workshop on Waldenström's Macroglobulinemia (IWWM). The study comprised an initial screening phase (up to 28 days), a single-arm treatment phase, and a follow-up phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical and definitive histologic diagnosis of WM, meeting at least one criterion for treatment according to consensus panel criteria from the Seventh IWWM.
2. WM pathology confirmation by central lab prior to study enrollment. Previous pathology report, concurrently with newly generated central lab report to be reviewed to support WM diagnosis.
3. Men and women ≥ 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Previously treated with a minimum of 1 prior line of standard chemotherapy-containing regimen (with completion of ≥ 2 continuous treatment cycles).
6. Documented failure to achieve at least minor response or documented disease progression after response to the most recent treatment regimen.
7. Neutrophils ≥ 0.75 x 10^9/L independent of growth factor support within 7 days of first dose.
8. Platelets ≥ 50 x 10^9/L, independent of growth factor support or transfusion within 7 days of first dose.
9. Hemoglobin ≥80 g/L, independent of erythropoietin (EPO) support or transfusion within 7 days of first dose of study drug.
10. Creatinine clearance of ≥ 30 mL/min (as estimated by the Cockcroft-Gault equation or estimated glomerular filtration rate [eGFR] from the Modification of Diet in Renal Disease [MDRD]).
11. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x upper limit of normal (ULN).
12. Bilirubin ≤ 2 x ULN (unless documented Gilbert's syndrome).
13. International normalized ratio ≤ 1.5 and activated partial thromboplastin time ≤ 1.5 x ULN. Participants with lupus anticoagulant or acquired von Willebrand disease due to WM may be enrolled after discussion with the medical monitor.
14. ECHO must demonstrate left ventricular ejection fraction (LVEF) ≥50%.
15. Participants who relapse after autologous stem cell transplant may be enrolled if they are at least 6 months after transplant at screening. To be eligible after transplant, participants should have no active related infections.
16. Females of childbearing potential must agree to use highly effective forms of birth control throughout the course of the study and at least up to 90 days after last dose of study drug. Highly effective forms of birth control can be defined as abstinence, hysterectomy, bilateral oophorectomy with no menstrual bleeding for up to 6 months, intrauterine contraception, hormonal methods such as contraceptive injection, oral contraceptive, etc. Males must have undergone sterilization-vasectomy, or use a barrier method where the female partner uses the effective forms of birth control noted above and must not donate sperm for at least 90 days after last dose of study drug.
17. Life expectancy of > 4 months.
18. Able to provide written informed consent and can understand and comply with the requirements of the study.

Key Exclusion Criteria:

1. Central nervous system (CNS) involvement by WM.
2. Prior exposure to a BTK inhibitor.
3. Evidence of disease transformation.
4. Prior corticosteroids given in excess of prednisone 10 mg/day or its equivalent with antineoplastic intent within 7 days, prior chemotherapy, targeted therapy, or radiation therapy within 3 weeks, antineoplastic therapy with Chinese herbal medicine or antibody based therapies within 4 weeks of the start of study drug.
5. Major surgery within 4 weeks of randomization.
6. Toxicity of ≥ Grade 1 from prior anti-cancer therapy (except for absolute neutrophil count [ANC], platelets, and hemoglobin. For ANC, platelets, and hemoglobin, please follow inclusion criteria #7 [neutrophils], #8 [platelets], and #9 [hemoglobin]).
7. History of other active malignancies within 2 years of study entry, with exception of (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent.
8. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any Class 3 or 4 cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification, or history of myocardial infarction within 6 months of screening.
9. QTcF prolongation (defined as a QTc >480 msecs based on Fridericia's formula) or other significant ECG abnormalities including second degree atrioventricular (AV) block Type II, or third degree AV block.
10. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
11. Active infection including infections requiring oral or intravenous anti-microbial therapy.
12. Known human immunodeficiency virus (HIV), or active hepatitis B or hepatitis C infection (detected positive by polymerase chain reaction [PCR]).
13. Pregnant or lactating women.
14. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study at risk.
15. On medications which are strong CYP3A inhibitors or strong CYP3A inducers.
16. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
17. Has received allogenic hematopoietic stem cell transplantation prior to enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (10):
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] An G, Zhou D, Cheng S, Zhou K, Li J, Zhou J, Xie L, Jin J, Zhong L, Yan L, Guo H, Du C, Zhong J, Yu Y, Wu B, Qiu L. A Phase II Trial of the Bruton Tyrosine-Kinase Inhibitor Zanubrutinib (BGB-3111) in Patients with Relapsed/Refractory Waldenstrom Macroglobulinemia. Clin Cancer Res. 2021 Oct 15;27(20):5492-5501. doi: 10.1158/1078-0432.CCR-21-0539. Epub 2021 Jul 12. PMID 34253577
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants at 10 study centers in China. The first participant was dosed on 31 August 2017, and the last participant enrolled and received their first dose of zanubrutinib on 08 May 2018. A total of 44 participants were enrolled and all received at least 1 dose of the study drug.
Pre-assignment Details: The protocol-defined efficacy analyses were performed 12 months after the last patient received the first dose of study drug, with a data cutoff date of 08 May 2019.
Period: Overall Study
Arm/Group | Zanubrutinib
Started | 44
Completed | 0
Not Completed | 44
Not completed — Death | 7
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2
Not completed — Transferred to long-term extension study | 29

BASELINE CHARACTERISTICS:
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 44

OUTCOME MEASURES:

1. Primary Outcome: Major Response Rate (MRR) as Assessed by the Independent Review Committee
Description: MRR is defined as the percentage of participants who achieved complete response (CR) + very good partial response (VGPR) + partial response (PR), as assessed by an independent review committee according to modified Owen's criteria
Time Frame: Up to approximately 1 year and 9 months
Population: Efficacy Analysis Set includes participants with confirmed Waldenström's macroglobulinemia based on central pathologic review among those who received at least one dose of study drug and with a baseline IgM (or M-protein) ≥ 5 g/L
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Percentage of participants | 69.8 [53.87 to 82.82]
Statistical Analysis 1: Comparison: Zanubrutinib; Zanubrutinib versus historical control estimate of 30%; Test type: Superiority; p < 0.0001, Exact binomial test — P value was based on the exact binomial test against the null hypothesis H0: MRR = 0.30 at a significance level of 0.025 (1-sided)

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by an independent review committee using modified Owen's criteria
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Months | NA [16.53 to NA] — NA = not estimable; could not be calculated due insufficient number participants with events

3. Secondary Outcome: PFS: Event-free Rate
Description: Progression/death event-free rates were estimated by Kaplan-Meier method with 95% confidence intervals (CIs) estimated using Greenwood's formula
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Percentage of participants
  6 months | 89.8 [75.1 to 96.1]
  9 months | 87.0 [71.5 to 94.4]
  12 months | 77.8 [60.2 to 88.3]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a minor, partial, very good partial, and complete response, as assessed by an independent review committee using modified Owen's criteria
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Percentage of participants | 79.1 [63.96 to 89.96]

5. Secondary Outcome: Duration of Major Response (DOMR)
Description: DOMR is defined as the time from the date that the major response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever comes first, as assessed by an independent review committee using modified Owen's criteria
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Months | NA [13.77 to NA] — NA = not estimable, could not be calculated due insufficient number participants with events

6. Secondary Outcome: DOMR: Event-free Rate
Description: DOMR event-free rates were estimated by Kaplan-Meier method with 95% CIs estimated using Greenwood's formula
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Percentage of participants
  6 months | 96.2 [75.7 to 99.4]
  9 months | 87.0 [64.7 to 95.6]
  12 months | 87.0 [64.7 to 95.6]

7. Secondary Outcome: Number of Participants With Resolution of Treatment-precipitating Symptoms
Description: Number of participants with resolution of treatment-precipitating symptoms, defined as any resolution (from "Yes" at baseline to "No" at any postbaseline point onwards during study) of the indications for initiation of therapy in WM signs and symptoms evaluation.
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Participants | 35

8. Secondary Outcome: Number of Participants With an Anti-lymphoma Effect
Description: Number of participants with an anti-lymphoma effect, defined as any reduction during the course of study in bone marrow involvement by lymphoplasmacytoid lymphocytes and/or size of lymphadenopathy and/or splenomegaly by computed tomography scan as assessed by an independent review committee; lymphadenopathy is defined as any node with longest diameter (LDi) > 1.5 cm and splenomegaly is defined as vertical spleen length > 13 cm
Time Frame: Up to approximately 1 year and 9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 43
Participants | 34

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs), grade 3 or higher TEAEs, serious adverse events (SAEs), treatment-related adverse events (AEs), adverse events of special interest, and TEAEs leading to study drug discontinuation, dose reduction and treatment interruption
Time Frame: Up to approximately 3 years and 5 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 44
Participants
  At least one TEAE | 44
  Grade 3 or higher TEAEs | 34
  Serious TEAEs | 25
  Treatment-related TEAEs | 41
  TEAEs of special interest | 43
  TEAEs leading to study drug discontinuation | 5
  TEAEs leading to treatment interruption | 17
  TEAEs leading to dose reduction | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years and 5 months
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event that had an onset or worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days after the last dose of study drug or initiation of new anticancer therapy, whichever occurred first. Worsening of an event to Grade 5 beyond 30 days after the last dose of study drug was also considered a TEAE (if prior to start of new anticancer therapy).
Arm/Group | Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 7/44
Serious Adverse Events (participants affected / at risk) | 25/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=44)
Anaemia (Blood and lymphatic system disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Dysbiosis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Abscess limb (Infections and infestations) | 1
Acute hepatitis B (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 10
Pulmonary mycosis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial mass (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=44)
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Cataract (Eye disorders) | 3
Conjunctival haemorrhage (Eye disorders) | 2
Ocular discomfort (Eye disorders) | 2
Retinal haemorrhage (Eye disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 11
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 5
Chest pain (General disorders) | 2
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 6
Bronchitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 6
Periodontitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 8
Fracture (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Bilirubin conjugated increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood immunoglobulin M increased (Investigations) | 2
Carbon dioxide increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 26
Platelet count decreased (Investigations) | 13
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 10
White blood cell count decreased (Investigations) | 14
White blood cells urine positive (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 7
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2
Neurodermatitis (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03332173/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03332173/SAP_001.pdf